CLINICAL TRIAL: NCT05001477
Title: Customized TULSA-PRO Ablation Registry
Acronym: CARE
Status: Recruiting | Type: Observational
Sponsor: Profound Medical Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: GCP-10250
Record Dates: First submitted 2021-05-13; First posted 2021-08-12 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2023-11

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma; Benign Prostatic Hyperplasia
Keywords: Prostate ablation; high intensity transurethral ultrasound ablation; MRI-guided; minimally invasive; real-time temperature feedback control; prostate cancer; BPH; TULSA
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 40 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: TULSA Procedure — Transurethral ultrasound ablation procedure

SUMMARY:
This patient registry will capture data from patients who have been or who are undergoing the transurethral ultrasound ablation (TULSA) procedure as part of their routine clinical care. The registry will shed light on real-world outcomes of safety and efficacy of the procedure and understand how a patient's quality of life is affected throughout their follow-up and lifetime.

DETAILED DESCRIPTION:
This registry will capture data on patients undergoing customized transurethral ultrasound ablation (TULSA) as part of their routine clinical care. The aim of collecting such data is to further evaluate real-world outcomes of safety and efficacy of this treatment. The collection of this data is intended to form an evidence-base from which conclusions can be drawn on how to optimize outcomes to improve patient care and QOL, and further expand on knowledge of practice trends and treatment costs.

The primary safety objective is to estimate the rate of complications attributable to the TULSA Procedure. The primary efficacy objective is estimating the proportion of patients who are free from primary treatment failure after the TULSA Procedure.

Patients being offered TULSA Procedure will be invited to participate in the registry. Patients who have already undergone TULSA will also be allowed to join the registry. Hundreds to thousands of patients across sites in US, Canada and Europe will be followed as per routine clinical care at 3 months, 6 months, 12 months, 2 years, 3 years, 4 years, 5 years and annually lifelong thereafter. Patients will remain active in the registry until they voluntarily withdraw or die. At each visit, patients will complete a set of questionnaires that is sent to them by email.

* Informed consent will be collected prior to enrolling the patient into the Registry.
* Initial baseline information will be collected (eg. demographics, medical history, concomitant medication, prostate MRI, prostate biopsy, PSA, and QOL Questionnaires)
* TULSA Procedure treatment assessment and complications will be collected from clinic records from treatment day. Optional financial tracking information may also be collected if patient consents to this portion of the registry.
* At follow-up visits, a set of data points will be collected (eg. PSA, complications, QoL Questionnaires, survival assessments, and optional financial tracking information)

All Registry data will be collected and stored in an electronic database capture system called Castor. Castor is validated and compliant with all applicable laws and regulations, including ICH E6 GCP, 21 CFR Part 11, EU annex II, General Data Protection Regulation (GDPR), HIPAA (US), ISO 9001 and ISO 27001. Only sites and sponsor personnel will have access to the database. On site and/or remote study monitoring will be undertaken to check source documents and accuracy of data entry. All reasonable methods will be used to try to minimize missing data, however, some missing data is expected to occur. No interpolation of missing data will occur. Standard descriptive statistics, including the mean, standard deviation, median, range, proportion and frequency, will be used throughout to summarize results. Measures will be presented, and 95% confidence intervals will be constructed for selected measures, such as efficacy and safety. As a primarily descriptive study, analyses will be performed at the p=0.05 level of significance and exact analyses will be used wherever possible.

ELIGIBILITY:
Inclusion Criteria

1. Male
2. >18 years old
3. Candidate for TULSA-PRO treatment
4. willing and able to sign the Informed Consent form

Exclusion Criteria:

None.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include as many eligible subjects as willing to participate who have undergone or will be undergoing the TULSA Procedure.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-10-27 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2061-10 (Estimated)

PRIMARY OUTCOMES:
Rate of complications | 5 years
  estimating the rate of complications (Clavien-Dindo grades III - IV) attributable to the TULSA Procedure
Freedom from treatment failure | 5 years
  Estimating the proportion of patients who are free from primary treatment failure after the TULSA Procedure.

SECONDARY OUTCOMES:
Complications Data | Lifelong up to 99 years
  complications arising from TULSA-PRO treatment, categorized based on the type of corrective therapy needed using the Clavien-Dindo classification system
Biopsy Data | Between 6 and 18 months post TULSA Procedure
  in men with prostate cancer, biopsy data to assess if there are changes to either cancer or clinically significant cancer in the treatment region.
Prostate Volume Reduction on MRI | Between 6 and 18 months post TULSA Procedure
  Multi-parametric prostate MRI data to measure prostate volume reduction
Suspicious cancerous lesions on MRI | Between 6 and 18 months post TULSA Procedure
  Identify presence of any suspicious (i.e. suspected for cancer) lesions.
PSA Data | Lifelong up to 99 years
  PSA data to identify changes in PSA from baseline.
QoL (IIEF-5) Data-Evaluation of Erectile Dysfunction, Ejaculatory function and erection firmness | Lifelong up to 99 years
  Patient-reported qualify of life (QoL) questionnaire answers to assess changes in erectile dysfunction, ejaculatory function and erection firmness:
  IIEF-5 (International Index of Erectile Function) Minimum score=5, Maximum score=25. Lower scores indicate a worse outcome.
QoL (IIEF-15) Data-Evaluation of Erectile Dysfunction, Ejaculatory function and erection firmness | Lifelong up to 99 years
  Patient-reported qualify of life (QoL) questionnaire answers to assess changes in erectile dysfunction, ejaculatory function and erection firmness.
  2 questions from IIEF-15 (International Index of Erectile Function) Low scores indicate a worse outcome.
QoL (IPSS) Data- Evaluation of Urinary Symptoms and Incontinence | Lifelong up to 99 years
  Patient-reported qualify of life (QoL) questionnaire answers to assess changes in urinary symptoms and urinary incontinence:
  IPSS (International Prostate Symptom Score) Minimum score=0, Maximum score=35. Higher scores indicate a worse outcome.
QoL (EPIC) Data- Evaluation of Urinary Symptoms and Incontinence | Lifelong up to 99 years
  Patient-reported qualify of life (QoL) questionnaire answers to assess changes in urinary symptoms and urinary incontinence:
  2 questions from EPIC-26 (Expanded Prostate Cancer Index Composite)
Survival Data- Percentage of participants without Biochemical Recurrence | Lifelong up to 99 years
  in men with prostate cancer, survival data will be captured to identify percentage of participants who are free from biochemical recurrence.
Survival Data- Percentage of participants without additional Salvage Treatment | Lifelong up to 99 years
  in men with prostate cancer, survival data will be captured to identify percentage of participants who are free from undergoing any additional salvage treatment.
Survival Data- Percentage of participants without additional Systemic Therapy | Lifelong up to 99 years
  in men with prostate cancer, survival data will be captured to identify percentage of participants who are free from undergoing any additional systemic therapy.
Survival Data- Percentage of participants without Distant Metastases | Lifelong up to 99 years
  in men with prostate cancer, survival data will be captured to identify percentage of participants who are free from distant metastases.
Survival Data- Number of patients with disease-specific mortality | Lifelong up to 99 years
  in men with prostate cancer, survival data will be captured to identify freedom from disease-specific mortality.
Survival Data- Overall mortality | Lifelong up to 99 years
  in men with prostate cancer, survival data will be captured to identify freedom from overall mortality.
Financial Data- Total Costs | Between 0 and 3 months post Tulsa Procedure
  Financial tracking information such total cost to patient, private insurance, public insurance) associated with treatment and visit will be collected.
Survival Data - Percentage of patients that got additional treatments for BPH | Lifelong up to 99 years
  Additional treatments related to urinary symptoms attributed to BPH will be collected, including types of treatments.
Survival Data - Dates of additional treatments undertaken for BPH patients | Lifelong up to 99 years
  Additional treatments related to urinary symptoms attributed to BPH will be collected, including dates of these treatments.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - RadNet's Liberty Pacific West Hills Facility, West Hills, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Wellspan Health, York, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Urology Place, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No